CLINICAL TRIAL: NCT06566235
Title: Cultural Adaptation and Implementation of Dialectical Behavior Therapy Skills Training Group for Adolescents With Emotional Disorders: a Feasibility Study and a Randomized Controlled Trial
Brief Title: Cultural Adaptation and Implementation of DBT for Adolescents With Emotional Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shen-Ing,Liu, Senior Attending Psychiatrist, Professor, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSTC 113-2314-B-195 -012 -MY3
Record Dates: First submitted 2024-08-10; First posted 2024-08-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-06

CONDITIONS: Emotional Disorders
Keywords: Dialectical Behavior Therapy Skills Training Group; Adolescents; Emotional Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally adapted DBT-A-ST group (Experimental): The culturally adapted DBT-A-ST consists of 15 weekly group sessions, each lasting 120 minutes, including a 10-minute break. It maintains the core elements of standard DBT-A, including its philosophical foundation and treatment strategies.
  Therapists focus on teaching DBT skills through various methods such as modeling, structured behavioral rehearsals, and feedback. Each session begins with a 40-minute group mindfulness exercise and homework review, followed by 60 minutes dedicated to skill-specific didactics and experiential activities, concluding with a 10-minute homework assignment. Two group leaders facilitate the sessions, and participants track their skill usage daily with diary cards, which are reviewed weekly.
  Interventions: Behavioral: Culturally adapted DBT-A-ST group
- Activities-based support group (ASG) (Placebo Comparator): ASG, based on principles of client-centered supportive therapy, is widely used by occupational therapists in mental health settings. ASG therapists aim to foster a sense of belongingness, maintain unconditional positive regard, and provide empathy, psychoeducation, and a treatment structure. Two group leaders held the sessions; teaching DBT skills and using cognitive behavioral strategies are prohibited. Each session starts with a review of their experiences over the last week (30 min), a support-building activity (30 min), and ends with an open group discussion about topics participants choose each week (50 min). For homework, participants will be asked to think about issues discussed and to track daily social support on diary cards.
  Interventions: Behavioral: Activities-based support group (ASG)

INTERVENTIONS:
Behavioral: Culturally adapted DBT-A-ST group — The culturally adapted DBT-A-ST consists of 15 weekly group sessions, each lasting 120 minutes, including a 10-minute break. It maintains the core elements of standard DBT-A, including its philosophical foundation and treatment strategies.
  Therapists focus on teaching DBT skills through various methods such as modeling, structured behavioral rehearsals, and feedback. Each session begins with a 40-minute group mindfulness exercise and homework review, followed by 60 minutes dedicated to skill-specific didactics and experiential activities, concluding with a 10-minute homework assignment. Two group leaders facilitate the sessions, and participants track their skill usage daily with diary cards, which are reviewed weekly.
  Arms: Culturally adapted DBT-A-ST group
Behavioral: Activities-based support group (ASG) — ASG, based on principles of client-centered supportive therapy, is widely used by occupational therapists in mental health settings. ASG therapists aim to foster a sense of belongingness, maintain unconditional positive regard, provide empathy, psychoeducational and a treatment structure. Two group leaders held the sessions, teaching DBT skills and using cognitive behavioral strategies are prohibited. Each session starts with a review of their experiences over the last week (30 min), a support-building activity (30 min), and ends with an open group discussion about topics participants choose each week (50 min). For homework, participants will be asked to think about issues discussed and to track daily social support on diary cards.
  Arms: Activities-based support group (ASG)

SUMMARY:
The goal of this study is to learn if Dialectical behavior therapy Skills

Training for Adolescents (DBT-A-ST) works on emotional disorders in adolescents. The main questions it aims to answer are:

Does DBT-A-ST produce faster improvements (i.e., steeper slopes), compared to ASG, on primary and secondary outcome measures during treatment and 3-month follow-up?

Does DBT-A-ST produce greater improvements, compared to ASG, on primary and secondary outcome measures?

Participants will:

Randomly assigned to (a) a culturally adapted DBT-A-ST or (b) activities-based support group (ASG).

Received five assessments before the start of the trial (T1), after 4, 8 sessions (T2, T3), at post-intervention (T4), and 3-month follow-up (T5).

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted in a medical center's child adolescent psychiatry department. Participants aged 12-17 years with current depressive or anxiety disorders as diagnosed using the K-SADS-E will be recruited and randomly allocated 1:1 to one of two study arms: a) culturally adapted DBT-A-ST group, b) Activities-based support group. Both interventions are in group format and include 15 weekly sessions, 120 min/each session. Based on power calculation, a target sample size of 160 youths will be included. Assessments will occur before the trial starts, at the 4th and 8th treatment sessions, in the end, and at the 3-month follow-up.

Primary outcomes are the severity of depression and anxiety, rated by blind assessors. Secondary outcomes include general psychopathology, number of DSM-5 disorders, quality of life, and self-reported measures. The treatment mechanisms and implementation processes will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years of age,
* informed consent is provided by the youth and one of the parents,
* Mandarin Chinese language proficiency sufficient to complete study questionnaire,
* a total score of either the PHQ-9≥ 10 or the GAD-7 ≥ 10,
* a current diagnosis of depressive or anxiety disorder from a K-SADS-E interview, including depression (F32-33); persistent mood disorder (F34), phobic anxiety disorder (F40), other anxiety disorder (F41), and adjustment disorders (F43.2).

Individuals with comorbid diagnoses of several emotional disorders are also enrolled. Comorbidities will not be stratified because this will significantly increase the complexity of the design (i.e., some patients may have multiple comorbid diagnoses).

Exclusion Criteria:

* diagnoses of intellectual disability, schizophrenia, pervasive developmental disorder, anorexia nervosa and substance use disorder in the past 3 months,
* active suicidal ideation with a plan or a history of frequent or recent suicide risk in the past 3 months,
* ADHD without elevations in the areas of anxiety, depression, or stress problems on the CBCL,
* recent (past 4 weeks) change in psychiatric medication or unwillingness to maintain a stable dosage of medication during study participation,
* had received five or more sessions of CBT in the past or unwilling to stop concurrent psychotherapy,
* any mental or physical condition requiring hospital admission,
* severe medical condition.

As we also aim for a naturalistic setting, we do not exclude patients who undergo medication changes during the trial if the treating clinician judges this to be necessary or clinically important.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale-17 item (HAMD-17) | baseline, 5-month and 8-month follow-up
  Hamilton Depression Scale-17 item (HAMD-17) is an outcome measure widely used in clinical.
  trials, with high score indicating a high degree of depression
Hamilton Anxiety Scale (HAM-A) | baseline, 5-month and 8-month follow-up
  Hamilton Anxiety Scale (HAM-A) comprises 14 items with each item being divided into five grades, based on a scale of 0 to 4. A high score indicates a high degree of anxiety.
Clinical Global Impressions-Severity (CGI-S) | baseline, 5-month and 8-month follow-up
  Clinical Global Impressions-Severity (CGI-S) is a standardized assessment tool used by clinicians to rate the severity of illness, change over time, and efficacy of medication.
Clinical Global Impressions-Improvement (CGI-I) | baseline,5-month and 8-month follow-up
  Clinical Global Impression-Improvement (CGI-I), is also a 7-point scale that assesses how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shen-Ing Liu, Ph.D, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No